CLINICAL TRIAL: NCT01418183
Title: Intra-operative Trigeminal Nerve Block For Post-operative Pain Control After Orthognathic Surgery
Brief Title: Pain Control After Orthognathic Surgery
Acronym: PCOGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100-0548A3
Record Dates: First submitted 2011-08-12; First posted 2011-08-17 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-06

CONDITIONS: Postoperative Pain
Keywords: Orthognathic surgery; Pain control; Trigeminal nerve; Levobupivacaine
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5ml 5% levobupivacaine (Experimental): 5ml 5% levobupivacaine to both maxillary and mandibular branches of trigeminal nerve on experimental side. (total 10ml)
  Interventions: Procedure: Trigeminal nerve block
- 5ml normal saline (Placebo Comparator): 5ml for maxillary and mandibular branches of trigeminal nerve (total 10ml on controlled side)
  Interventions: Procedure: Trigeminal nerve block
- 2.5ml 5% levobupivacaine (Experimental): 2.5ml 5% levobupivacaine to both maxillary and mandibular branches of trigeminal nerve on experimental side. (total 10ml)
  Interventions: Procedure: Trigeminal nerve block

INTERVENTIONS:
Procedure: Trigeminal nerve block — 5ml of long-effective local analgesics (5% levobupivacaine) will be delivered to maxillary and mandibular branches of trigeminal nerve.
  Other Names: 5ml Chirocaine
  Arms: 5ml 5% levobupivacaine
Procedure: Trigeminal nerve block — 2.5ml of long-effective local analgesics (5% levobupivacaine) will be delivered to maxillary and mandibular branches of trigeminal nerve.
  Other Names: 2.5ml Chirocaine
  Arms: 2.5ml 5% levobupivacaine
Procedure: Trigeminal nerve block — 5ml Normal saline will be delivered to maxillary and mandibular branches of trigeminal nerve.
  Other Names: Placebo
  Arms: 5ml normal saline

SUMMARY:
This study will assess the efficacy and safety of levobupivacaine for postoperative pain control in patients received orthognathic surgery. In this split-mouth study, each side will be randomized to receive 1) 5ml 0.5% levobupivacine, 2) 2.5ml 0.5% levobupivacaine, or 3) placebo. One shot of these agents will be delivered by nerve block to maxillary and mandibular branches of trigeminal nerve before the incision was made. The degree of postoperative pain will be evaluated daily by visual analog scale for up to 3 days. The anticipated time on study is 1 year, and the target sample size is 40 individuals.

DETAILED DESCRIPTION:
Design of intervention vs. control Intra-operative injective of (chirocaine) before incision Location of injection: inferior alveolar nerve proximal to its entrance to ramus of mandible, maxillary nerve around pterygopalatine ganglion Amount of injection on each injection site: (1) Experimental group 1: 5mg/ml chirocaine 5cc (2)Experimental group 2: 5mg/ml chirocaine 2.5cc (3)Control group: normal saline 5cc. There are totally 4 injection sites for two jaw surgery and 2 injection sites for one jaw surgery. The experimental site and control site will be determined randomly before injection.

Outcome measurement

* Primary: effectiveness of intra-operative nerve block on post-operative pain control
* Secondary:

  1. whether the pain relieve effect is dose-related
  2. how long will this effect last

The intensity of post-operative pain will be measured by VAS, visual analog scale)daily until patients are discharged.

Report adverse outcome:

* Intolerable pain on control group
* Adverse reaction to local anesthetic agent
* Injection-related complications (puncture of major vessels, hematoma on -injection site, etc.)

ELIGIBILITY:
Inclusion Criteria:

* all patients who will receive orthognathic surgery (one jaw or two jaw, with or without genioplasty) in Chang Gung Memorial Hospital since July 2011

Exclusion Criteria:

* more complex (2- or more piece LeFort I osteotomy, combined gonial resection in BSSO, etc.) or less complex (only Wassmund and/or Kole osteotomies in upper or lower jaw) orthognathic procedures
* unexpected fracture (unilateral)
* intra-operative nerve injuries
* significant facial asymmetry which demands different procedures (location of osteotomy, extension of muscle stripping, etc.)
* cleft patient, post-traumatic patients, patients with craniofacial syndromes or other neurological or systemic problems which might interfere pain evaluation post-operatively

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | participants will be followed for the duration of hospital stay, an expected average of 3days
  The degree of pain will be measured daily by visual analog scale.

SECONDARY OUTCOMES:
Effective duration of levobupivacaine nerve block | participants will be followed for the duration of hospital stay, an expected average of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chieh Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan